CLINICAL TRIAL: NCT04486807
Title: Shoulder Muscle Imbalance as a Risk Factor for Shoulder Injury in Elite Adolescent Badminton Players: a Prospective Pilot Study
Brief Title: Shoulder Muscle Imbalance as a Risk Factor for Shoulder Injury in Elite Badminton Players
Acronym: BADEPAULE
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Joffrey DRIGNY, Principal Investigator, Chief Resident in the Sport Medicine Department (MD), PhD student, University Hospital, Caen
Other Study IDs: BADEPAULE
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Sport Injury; Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Elite badminton players — The population was all the elite badminton players followed in a University Hospital Centre and the National Institute of Sport, Expertise, and Performance. We excluded players who had SSI in the 3 months prior to the isokinetic test or had shoulder surgery. They were included and followed during the badminton season (Nineteen elite badminton players and followed over the badminton season (from september 2018 to may 2019 or from september 2019 to may 2020)

SUMMARY:
Background: To assess the impact of pre-season clinical measures and rotator muscles strength on the risk of significant shoulder injury (SSI) in elite badminton players Design: Prospective cohort study Participants: Nineteen elite adolescents badminton players were included and followed over the badminton season (from september 2018 to may 2019 and/or from september 2019 to may 2020) .

Independent variables: A pre-season visit consisted in clinical and isokinetic shoulder strength testing. Clinical testing consisted in the shoulder range of motion (ROM) measurements and the table-to-acromion distance (TAD)Isokinetic internal and external rotator shoulder muscles strength was tested at 60 and 240°/s. Conventional and functional (eccentric-to-concentric) ratios (FR) were calculated. SSI collection was performed by an experienced sport physician.

ELIGIBILITY:
Inclusion Criteria:

All the elite badminton players from a high-level club and the National Institute of Sport, Expertise, and Performance

Exclusion Criteria:

Players who had SSI in the 3 months prior to the isokinetic test or had shoulder surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nineteen elite badminton players and followed over the badminton season (from september 2018 to may 2019 or from september 2019 to may 2020)
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Baseline Isokinetic strength testing (peak torques) | one preseason evaluation (september 2018 or september 2019)
  Shoulder rotator muscles isokinetic strength test, Measures: Peak Torque on internal rotator muscles (IR) and external rotator muscles (ER), in NM (newton.meter)
Baseline Isokinetic strength testing (ratios) | one preseason evaluation (september 2018 or september 2019)
  Shoulder rotator muscles isokinetic strength test, Measures: ratios between external rotator muscles (ER) and internal rotator muscles (IR) (ER:IR), in percent (%)
Clinical measurements, ROM | ne evaluation, one preseason visit (september 2018 or september 2019)
  Shoulder internal and external rotation range of motion (ROM)
Clinical measurements TAD | one preseason visit (september 2018 or september 2019)
  table-to-acromion distance (in cm)
Significant Shoulder Injury (SSI) collection (number of injury) | During the badminton season, the number (number, n) of injury was recorded from september 2018 to may 2019 or from september 2019 to may 2020
  Significant Shoulder Injury (SSI) collection for the number of injury
Significant Shoulder Injury (SSI) collection (type of injury) | During the badminton season, the type of injury (number, n) was recorded from september 2018 to may 2019 or from september 2019 to may 2020
  Significant Shoulder Injury (SSI) collection for the type of injury
Significant Shoulder Injury (SSI) collection (time lost from participation) | During the badminton season, the time lost from participation was recorded (in days) from september 2018 to may 2019 or from september 2019 to may 2020
  Significant Shoulder Injury (SSI) collection for time lost from participation due to the injury

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France